CLINICAL TRIAL: NCT07365995
Title: A Phase III, Randomized, Open-label Trial of BNT324 Versus Docetaxel With Prednisone/Prednisolone in Metastatic Castration-resistant Prostate Cancer
Brief Title: A Phase III Trial of BNT324 Versus Docetaxel in Metastatic Castration-resistant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: BioNTech Shanghai Pharmaceutical Co., Ltd. (Unknown); DualityBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT324-03; 2025-524445-27-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-23; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Immunotherapy; Antibody-drug conjugate (ADC); Standard of care (SoC); Chemotherapy; Steroids; BNT324 (DB-1311); mCRPC
MeSH Terms: interventions — Docetaxel; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNT324 (Experimental)
  Interventions: Drug: BNT324
- Docetaxel plus prednisone/ prednisolone (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: Prednisone/prednisolone

INTERVENTIONS:
Drug: BNT324 — Intravenous infusion
  Other Names: DB-1311
  Arms: BNT324
Drug: Docetaxel — Intravenous infusion
  Arms: Docetaxel plus prednisone/ prednisolone
Drug: Prednisone/prednisolone — Oral
  Arms: Docetaxel plus prednisone/ prednisolone

SUMMARY:
This study will test whether BNT324 is safe and works better against metastatic castration-resistant prostate cancer (mCRPC) than the current standard of care (SoC) chemotherapy, which is docetaxel (given together with the steroid medicines prednisone or prednisolone). The study will include participants with mCRPC that have been previously treated with androgen receptor pathway inhibitor, but with no previous taxane-based systematic chemotherapy for mCRPC.

The main goals of this study are:

* To find out if BNT324 helps participants live longer without their cancer getting worse (radiographic progression-free survival [rPFS]).
* To find out if BNT324 helps participants live longer overall (overall survival [OS]).

DETAILED DESCRIPTION:
The study consists of a screening period (up to 28 days), a treatment period with 21-day cycles, and an after-treatment period that includes a 30-day safety follow-up period and a long-term survival follow-up period.

Treatment continues until the cancer clearly gets worse (in scans, based on blinded independent central review [BICR] assessment or investigator's decision), side effects become unacceptable, the participant chooses to stop, or the study ends.

Participants are put into one of two groups in a 1:1 ratio, which means they will have an equal chance to be in either treatment group, i.e., BNT324 group, or docetaxel plus prednisone/prednisolone group (current SoC). An independent committee will help ensure participant safety, by regularly reviewing safety and early results.

For each participant, the treatment and follow-up periods are projected to be up to ~58 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Are male adults (defined as ≥18 years of age or of an acceptable age according to local regulations at the time of giving informed consent).
* Must have documented progressive prostate cancer based on at least one of the following criteria:

  * Serum/plasma PSA progression, by local laboratory, defined as two consecutive increases in PSA over a previous reference value, each measured sequentially at least 1 week apart. The PSA value at screening is required to be ≥1.0 ng/mL.
  * Radiographic soft tissue progression as per PCWG3-modified RECIST v1.1.
  * Radiographic progression of bone disease: evaluable disease or new bone lesion(s) by bone scan per PCWG3 criteria.
* Had previously received one or two prior androgen receptor pathway inhibitor treatments and experienced disease progression during or after a minimum of 8 weeks of therapy.
* Must not have received systemic cytotoxic chemotherapy, including taxane-based chemotherapy, for mCRPC.
* Must have had prior orchiectomy and/or have ongoing androgen-deprivation therapy and a castrate-level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L). Participant being treated with luteinizing hormone-releasing hormone agonists or antagonists must continue such treatment throughout the study.
* Must have an Eastern Cooperative Oncology Group performance score of 0 or 1.

Key Exclusion Criteria:

* Have received prior treatment with B7-H3 targeted therapy, including B7-H3 ADCs.
* Have uncontrolled or significant cardiovascular disease, as defined in the protocol.
* Have a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids or have current ILD/pneumonitis.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
rPFS assessed by BICR | From randomization to end of study, i.e., up to 58 months
  By arm. rPFS is defined as time from randomization to radiographic disease progression per Prostate Cancer Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria, or death from any cause, whichever occurs first.
OS | From randomization to end of study, i.e., up to 58 months
  By arm. OS is defined as time from randomization to death from any cause.

SECONDARY OUTCOMES:
Time to first subsequent therapy (TFTS) | From randomization to end of study, i.e., up to 58 months
  By arm. TFST is defined as time from randomization to initiation of the first subsequent systemic anticancer therapy or death, whichever occurs first.
Objective response rate (ORR) | From randomization to end of study, i.e., up to 58 months
  By arm. ORR is defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (per PCWG3-modifed RECIST v1.1 as assessed by BICR) is observed as best overall response.
Duration of response (DOR) | From randomization to end of study, i.e., up to 58 months
  By arm. DOR is defined as time from first objective response (confirmed CR or PR per PCWG3-modified RECIST v1.1 criteria as assessed by BICR) to first occurrence of objective tumor progression (progressive disease per PCWG3-modified RECIST v1.1 criteria as assessed by BICR) or death from any cause, whichever occurs first.
Time to pain progression (TTPP) | From randomization to safety follow-up visit (30 days after the last dose), i.e., up to 58 months
  By arm. TTPP is defined as time from randomization to pain progression as determined by Brief Pain Inventory-Short Form Item 3 "worst pain in 24 hours" and opiate analgesic use (Analgesic Quantification Algorithm score).
rPFS as assessed by investigator | From randomization to end of study, i.e., up to 58 months
  By arm. rPFS is defined as time from randomization to radiographic disease progression per PCWG3-modified RECIST v1.1 criteria, or death from any cause, whichever occurs first.
Time to first symptomatic skeletal-related event (SSRE) | From randomization to end of study, i.e., up to 58 months
  By arm. Time to first SSRE is defined as time from randomization to first occurrence of any of the following SSREs:
  * Use of external beam radiation therapy to prevent or relieve skeletal symptoms.
  * New symptomatic pathologic bone fracture (vertebral or non-vertebral).
  * Spinal cord compression.
  * Tumor-related orthopedic surgical intervention.
Time to prostate-specific antigen (PSA) progression (by central lab testing results) | From baseline to end of treatment visit, i.e., up to 58 months
  By arm. Time to PSA progression is defined as time from randomization to PSA progression per PCWG3 criteria.
PSA response (by central lab testing results) | From baseline to end of treatment visit, i.e., up to 58 months
  By arm. PSA response is defined as having a post-baseline PSA reduction ≥50% from baseline with a consecutive confirmation assessment at least 3 weeks later per PCWG3 criteria.
Number and percentage of participants with treatment-emergent adverse events (TEAEs) including Grade ≥3, serious, and fatal TEAEs | From the start of study treatment until 30 days after the last dose of study treatment or until start of new systemic anticancer therapy, whichever occurs first, i.e., up to 58 months
  TEAEs by relationship and by arm.
Number and percentage of participants with dose interruptions, reductions or discontinuations of study treatment due to TEAEs | From the start of study treatment until 30 days after the last dose of study treatment or until start of new systemic anticancer therapy, whichever occurs first, i.e., up to 58 months
  By arm.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE

IPD SHARING:
Plan to Share IPD: No